CLINICAL TRIAL: NCT05621889
Title: Impacts of an Innovative Patient-partner-guided Virtual Group Speech Pathology Intervention Model to Prevent Swallowing Disorders in Patients Treated With Chemoradiotherapy for Head and Neck Cancer
Brief Title: Innovative Patient-partner-guided Virtual Group Speech Pathology Intervention Model in Head and Neck Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Université du Québec à Trois-Rivières (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-11195
Record Dates: First submitted 2022-11-11; First posted 2022-11-18 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- virtual group speech therapy intervention guided by a patient partner (Experimental)
  Interventions: Procedure: virtual group speech therapy intervention guided by a patient partner

INTERVENTIONS:
Procedure: virtual group speech therapy intervention guided by a patient partner — virtual group speech therapy intervention guided by a patient partner

SUMMARY:
This project aims to study an innovative intervention, the eG2 Intervention, developed by speech-language pathologists at the Centre hospitalier de l'Université de Montréal to improve therapeutic adherence and prevent dysphagia in patients treated with chemoradiotherapy for head and neck cancer.

The innovation consists in offering a speech therapy intervention that is 1) virtual, 2) group-based (whereas it is usually individual) and 3) involves a patient partner. This intervention has the potential to improve quality of care, accessibility to services and optimize health care resources.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age with a diagnosis of head or neck cancer
* Chemoradiotherapy treatments planned for curative purposes
* Planned external radiation therapy dose of at least ≥60 Grays
* Sufficient proficiency in French to complete self-reported questionnaires

Exclusion Criteria:

* Remote metastases
* Previous or planned total laryngectomy
* Previous moderate/severe dysphagia known and/or evaluated by speech therapy
* Diagnosis of a second synchronous cancer at the time of study enrollment
* History of prior radiation therapy to the head and neck area
* Have a cognitive impairment (diagnosed or suspected) that may significantly interfere with participation in the intervention and various measurement procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Rate of nasogastric tube | within 6 weeks post radiation
  To evaluate the rate of nasogastric tube placement in the acute and subacute period in patients who participated in the group intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No